CLINICAL TRIAL: NCT05790512
Title: Association of Oral Helicobacter Pylori Infection With Gastric Helicobacter Pylori Infection
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232027-C-1-A
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Helicobacter Pylori
Keywords: Oral Helicobacter Pylori; Helicobacter Pylori Gastric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Both gastric and oral Helicobacter pylori are negative
- Negative for Helicobacter pylori for gastric and positive for Helicobacter pylori for oral cavity
- Positive for Helicobacter pylori for gastric and negative for Helicobacter pylori for oral cavity
- Both gastric and oral Helicobacter pylori are positive

SUMMARY:
The aim of this study was to investigate the association between oral Helicobacter pylori infection and gastric Helicobacter pylori infection. Patients who were tested for gastric Helicobacter pylori were tested for oral Helicobacter pylori at the same time, and were divided into four groups according to the test results to compare the positive rate of oral Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70 ,both gender.
2. Initial diagnosis of stomach Helicobacter pylori infection or never had Helicobacter pylori infection.
3. Have not received dental care or systemic periodontal basic treatment in the past 1 year.

Exclusion Criteria:

1. There is serious organ damage and complications (such as cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases.
2. Ongoing use of antiulcer medications (including PPIs taken within 2 weeks before Helicobacter pylori infection testing), antibiotics, or bismuth complexes (more than 3 times/week before screening).
3. Those with severe oral diseases and malignant tumors of the mouth.
4. Previously had upper gastrointestinal surgery.
5. Refusal to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients are from Xijing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Positive rate of oral Helicobacter pylori | 7 months
  The oral Helicobacter pylori test is performed using the Helicobacter pylori test kit

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China